CLINICAL TRIAL: NCT05547399
Title: A Single-dose, Open-label, Randomized, Crossover Study in Healthy Adult Subjects to Assess the Relative Bioavailability of a Zanubrutinib Tablet Compared to Zanubrutinib Capsules and to Evaluate the Effects of Food on the Pharmacokinetics of the Zanubrutinib Tablet
Brief Title: Relative Bioavailability of Zanubrutinib Tablets Compared to Capsules and Effects of Food on the Pharmacokinetics of the Tablet in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BGB-3111-115
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dose Cohort (Experimental): Zanubrutinib will be administered as a single low dose of treatment (tablet) or reference (capsule) on separate occasions across several treatment sequences
  Interventions: Drug: Zanubrutinib
- High Dose Cohort (Experimental): Zanubrutinib will be administered as a single high dose of treatment (tablet) or reference (capsule) on separate occasions across several treatment sequences
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Administered orally as a tablet or capsule
  Other Names: BGB-3111; Brukinsa

SUMMARY:
Study to assess the relative bioavailability of zanubrutinib tablets compared to capsules and to evaluate the effects of food on the pharmacokinetics (PK) of the zanubrutinib tablet.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kg/m^2, inclusive
* In good health, determined by no clinically significant findings from medical history, 12-lead ECGs, vital signs measurements, and clinical laboratory evaluations as assessed by the investigator or designee
* Female participants of non-childbearing potential only

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator or designee
* Evidence of any infections (bacterial, viral, fungal, parasitic) within 4 weeks prior to the first dose of study drug, as determined by the investigator or designee
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator or designee
* History or presence of an abnormal ECG prior to the first dose of the study drug that, in the opinion of the investigator or designee, is clinically significant
* Use or intent to use prescription medications within 14 days prior to dosing or nonprescription medications/products/supplements within 7 days prior to check-in
* Use of tobacco or nicotine containing products within 3 months prior to check-in

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC0-inf) | Predose and up to 48 hours postdose up to Day 7
Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC0-t) | Predose and up to 48 hours postdose up to Day 7
Maximum observed plasma concentration (Cmax) | Predose and up to 48 hours postdose up to Day 7
Time of the maximum observed plasma concentration (Tmax) | Predose and up to 48 hours postdose up to Day 7
Apparent terminal elimination half-life (t1/2) | Predose and up to 48 hours postdose up to Day 7
Apparent volume of distribution (Vz/F) | Predose and up to 48 hours postdose up to Day 7
Rate of decrease of concentration in the terminal phase (λz) | Predose and up to 48 hours postdose up to Day 7
Apparent oral clearance (CL/F) | Predose and up to 48 hours postdose up to Day 7

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to approximately 6 months
Number of participants with clinically significant laboratory values | Up to approximately 6 months
  Laboratory values are based on hematology, clinical chemistry, and urinalysis test results
Number of participants with clinically significant electrocardiogram (ECG) results | Up to approximately 6 months
Number of participants with clinically significant vital sign measurements | Up to approximately 6 months
  Vital sign measurements include supine blood pressure, supine pulse rate, respiratory rate, and oral body temperature

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (1):
- Fortrea Clinical Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes